CLINICAL TRIAL: NCT04311827
Title: The Effect of the Serratus Anterior Plane Block in Improving Pain and Respiratory Function in Trauma Patients Presenting to the Emergency Department With Multiple Rib Fractures.
Brief Title: Serratus Anterior Plane Block for Improving Pain and Respiratory Function in Patients With Multiple Rib Fractures
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Society for Academic Emergency Medicine (Other)
Responsible Party: Principal Investigator, Youyou Duanmu, Clinical Assistant Professor, Stanford University
Other Study IDs: 52801
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Rib Fracture Multiple

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Serratus anterior plane block and traditional analgesia: Serratus anterior plane block (Bupivacaine 75mg injected into facial plane once) Acetaminophen 1000mg IV every 6 hours as needed Toradol 15mg IV every 6 hours as needed Morphine 4mg every 2 hours as needed Hydromorphone 0.5mg IV every 2 hours as needed
  Interventions: Other: Serratus Anterior Plane Block
- Traditional analgesia: Serratus anterior plane block (Bupivacaine 75mg injected into facial plane once) Acetaminophen 1000mg IV every 6 hours as needed Toradol 15mg IV every 6 hours as needed Morphine 4mg every 2 hours as needed Hydromorphone 0.5mg IV every 2 hours as needed

INTERVENTIONS:
Other: Serratus Anterior Plane Block — Injection of bupivacaine 75mg above the serratus anterior facial plane in the anterior axillary line
  Groups: Serratus anterior plane block and traditional analgesia

SUMMARY:
This is an observational study which will evaluate the efficacy of the serratus anterior plane block for treating pain and respiratory capacity in patients with multiple rib fractures. When resources are available for a SAPB to be performed, patients will receive this block in addition to traditional pain medications, while at other times, patients will receive traditional pain medications only.

DETAILED DESCRIPTION:
Pain management by systemic analgesics and by nerve blocks are both standard of care and used in Emergency Department (ED) depending on the resources available. Not all ED physicians are trained or comfortable with the serratus anterior nerve block and thus it is not always available to patients and is provider dependent.

This is an observational study where patients with multiple rib fractures will receive either a serratus anterior plane block (SAPB) in addition to traditional forms of pain control when providers trained to perform the block are available, or will receive traditional forms pain control if trained personnel are not available. In addition to the serratus anterior plane block, standard forms of pain control in the Stanford Emergency Department include: oral or parenteral acetaminophen, oral or parenteral NSAIDs, oral or parenteral opiates, parenteral lidocaine, and parenteral ketamine.

Retrospective evaluation of the allocation of patients to either nerve block or no nerve block will be dictated by physician ability, time and resources to do the block. The efficacy of the block will be evaluated by serial measurements of pain score and respiratory capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 18 years of age
2. Presentation to Stanford University Hospital Emergency Department within 12 hours of a traumatic incident
3. Three or more anterior and/or lateral unilateral rib fractures diagnosed by CT
4. GCS 15, with the ability to discern and describe pain from rib fractures and give consent
5. Presentation to the Emergency Department between 7am and 11pm (for identification by research assistants)

Exclusion Criteria:

1. Posterior rib fractures
2. Bilateral rib fractures
3. Sternal fracture
4. Known allergy to local anesthetics
5. Pregnancy
6. Significant coagulopathy
7. Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients who are 18 years and older (of all genders and ethnic backgrounds) presenting to the Stanford University Emergency Department with multiple, acute, unilateral, antero-lateral rib fractures who meet inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in pain score | Before and 3 hours after analgesia administration
  Patient reported pain score from 0-10 (0 - no pain, 10 = worst pain imaginable).
Change in incentive spirometry volume | Before and 3 hours after analgesia administration
  Maximum inspiratory respiratory volume (measured in ml) recorded on single use of incentive spirometer device

SECONDARY OUTCOMES:
Analgesia administration | Up to 3 days
  Dosage of analgesic medications administered for pain during ED visit and hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Youyou Duanmu, MD, MPH, Principal Investigator — STANFORD HOSPITAL
Locations (1):
- Stanford University Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luftig J, Mantuani D, Herring AA, Dixon B, Clattenburg E, Nagdev A. Successful emergency pain control for posterior rib fractures with ultrasound-guided erector spinae plane block. Am J Emerg Med. 2018 Aug;36(8):1391-1396. doi: 10.1016/j.ajem.2017.12.060. Epub 2017 Dec 28. PMID 29301653
- [Background] Battle CE, Hutchings H, Evans PA. Risk factors that predict mortality in patients with blunt chest wall trauma: a systematic review and meta-analysis. Injury. 2012 Jan;43(1):8-17. doi: 10.1016/j.injury.2011.01.004. Epub 2011 Jan 22. PMID 21256488
- [Background] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Ho AM, Karmakar MK, Critchley LA. Acute pain management of patients with multiple fractured ribs: a focus on regional techniques. Curr Opin Crit Care. 2011 Aug;17(4):323-7. doi: 10.1097/MCC.0b013e328348bf6f. PMID 21716105
- [Background] Thiruvenkatarajan V, Cruz Eng H, Adhikary SD. An update on regional analgesia for rib fractures. Curr Opin Anaesthesiol. 2018 Oct;31(5):601-607. doi: 10.1097/ACO.0000000000000637. PMID 30020155
- [Background] Adhikary SD, Liu WM, Fuller E, Cruz-Eng H, Chin KJ. The effect of erector spinae plane block on respiratory and analgesic outcomes in multiple rib fractures: a retrospective cohort study. Anaesthesia. 2019 May;74(5):585-593. doi: 10.1111/anae.14579. Epub 2019 Feb 10. PMID 30740657
- [Background] Durant E, Dixon B, Luftig J, Mantuani D, Herring A. Ultrasound-guided serratus plane block for ED rib fracture pain control. Am J Emerg Med. 2017 Jan;35(1):197.e3-197.e6. doi: 10.1016/j.ajem.2016.07.021. Epub 2016 Jul 19. No abstract available. PMID 27595172
- [Background] Todd SR, McNally MM, Holcomb JB, Kozar RA, Kao LS, Gonzalez EA, Cocanour CS, Vercruysse GA, Lygas MH, Brasseaux BK, Moore FA. A multidisciplinary clinical pathway decreases rib fracture-associated infectious morbidity and mortality in high-risk trauma patients. Am J Surg. 2006 Dec;192(6):806-11. doi: 10.1016/j.amjsurg.2006.08.048. PMID 17161098
- [Background] Martin TJ, Eltorai AS, Dunn R, Varone A, Joyce MF, Kheirbek T, Adams C Jr, Daniels AH, Eltorai AEM. Clinical management of rib fractures and methods for prevention of pulmonary complications: A review. Injury. 2019 Jun;50(6):1159-1165. doi: 10.1016/j.injury.2019.04.020. Epub 2019 Apr 22. PMID 31047683